CLINICAL TRIAL: NCT01519622
Title: Impact of Disease on the Concept of End-of-life Decisions of the Elderly in the Community
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: K202/2011
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Last update posted 2012-01-27 (Estimated); Status verified 2012-01

CONDITIONS: Sick Elderly
Keywords: End of life decisions; Perception of illness
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sick elderly in community
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire to be distributed among sick elderly in the community

SUMMARY:
The purpose of this study is to determine the priorities of the elderly in the community about end-of-life decisions. To check the perception of the disease in the elderly in the community.

DETAILED DESCRIPTION:
This study is descriptive adapters which examines the relationship between illness perception and preferences of end of life decisions in the elderly in the community.

Population and sample: The target population will be elderly and healthy community elderly population was accessible due to a special branch of the club together in the center of the country. Sample to be a sample of convenience. The study will include 88 seniors aged 65 and over to get the power of 0.80 and alfa 0.05, Tools: The study used three tools.

* The first tool is a questionnaire on demographic and clinical details
* The second tool questionnaire the Long term support program (LTSP)
* The third tool is a questionnaire perception of the disease Revised Illness Perceptions Questionnaire (IPQR)

The research process:

Investigator will present the proposal to the Commissioner Fund hospitals and request approval for the study. After receiving approval from the director Department of Health fund the hospital will make data collection phase HMO, days and hours of reception. Interrogator he is to partition the questionnaires and will be present when filling out the questionnaires to help, if and created a situation of lack of understanding of the questionnaires. Scholar, came to the population for the Disabled arriving at the clinic visit, and introduce himself and the subject of research. investigator will indicate questionnaire is anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Chronic illness
* Literate in Hebrew
* Treated in community HMO

Exclusion Criteria:

* Someone hospitalized in previous year
* History of mental illness
* Cognitive problems

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Sick Elderly in the Community | One year
  Questionnaires regarding end-of-life decisions and perception of illness

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel